CLINICAL TRIAL: NCT05463484
Title: Effects of a Composition Delivered Via Toothpaste on the Oral Microbiome, pH, Nitrite/Nitrate Ratio, Elastases, and Inflammation in Patients With Oral Dysbiosis: A Controlled, Randomized, Double-blind Study. Part of Stop Dysbiosis Project
Brief Title: Effects of a Composition on the Oral Microbiome, pH, Nitrite/Nitrate Ratio, Elastases and Inflammation in Oral Dysbiosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mucosa Innovations, S.L. (Industry)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 02-2021
Record Dates: First submitted 2022-07-07; First posted 2022-07-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Oral Dysbiosis
Keywords: Gum inflammation; Periodontal Dysbiosis; Oral Dysbiosis
MeSH Terms: conditions — Gingivitis | interventions — Betaine; Xylitol

STUDY DESIGN:
Intervention Model Description: Three toothpastes will be included in the study; one with the composition including an olive product, betaine and xylitol, one with the same composition but without the olive product, betaine and xylitol, and one of a product marketed for gingivitis with and antimicrobial ingredient.
  Subjects are randomnly assigned and products will have a white label so that nor subject nor researcher will know the composition to be tested.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (Experimental): Toothpaste including an olive product, betaine and xylitol (Saliactive®).
  Interventions: Drug: Test composition Saliactive® (olive product, betaine and xylitol)
- Placebo product (Placebo Comparator): Toothpaste with the same composition as the test product but without olive product, betaine and xylitol.
  Interventions: Drug: Placebo
- Control product (Active Comparator): Toothpaste marketed for gingivitis with zinc mineral with antimicrobial activity.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Test composition Saliactive® (olive product, betaine and xylitol) — Fluoridated toothpaste with Saliactive®.
  Other Names: Saliactive®
  Arms: Test product
Drug: Placebo — Fluoridated toothpaste without Saliactive®.
  Other Names: Placebo fluoridated toothpaste without the test composition
  Arms: Placebo product
Drug: Control — Commercial Fluoridated toothpaste for gingivitis with zinc citrate.
  Other Names: Control commercial Fluoridated toothpaste for gingivitis with zinc citrate.
  Arms: Control product

SUMMARY:
Dysbiosis is a condition in which the normal function of an ecological net is altered. In dysbiosis a state of inflammation, a loss of hydration, a change in pH, a loss of the barrier function are all allies of key pathogens that initiate invasion and cytokine and pro-inflammatory mediators release that target other tissues and organs resulting in chronic inflammatory conditions.

In health there is a cross-talk between the host and the microbiota in order to maintain and promote a state of eubiosis with a local and general health gain. Dysbiosis reversion has not been solved with the use of antibacterials, antiseptics nor antibiotics.

Stop dysbiosis project is focussed on different aspects of human dysbiosis such as oral dysbiosis, skin dysbiosis, vaginal dysbiosis and cancer dysbiosis, between others including the current prospective interventional double-blind randomised clinical trial.

One of the most common oral dysbiosis is periodontal and mucosa dysbiosis that courses with inflammation of the gingiva (gingivitis). This inflammation induces specific enzymes that in a later stage destroy connective tissue. The current clinical trial analyzes the effect of a composition (Saliactive ®) delivered to the oral cavity via a daily use toothpaste (YOTUEL® microbiome toothpaste) in a group of patients with oral dysbiosis.

DETAILED DESCRIPTION:
Oral microbiota is the most diverse of the human body. It consists of mainly commensal bacteria, archea, protozoos, yeast and funghi. More than 700 species of bacteria have been identified in the mouth. In conditions of health these bacteria live in equilibrium. In inflammatory conditions, balance is lost, due to changes in microbiota or in the ecosystem with lost of the mucosa barrier function. If dysbiosis appears pathogen or fragments of these or toxic agents penetrate the body orchestrating a deep alteration of vital functions such as immune defense, nitric oxide pathways, cell cycle regulation and redox balance.

Periodontal dysbiosis is the consequence of the accumulation of plaque and the increase of gram negative species capable of releasing virulence factors that maintain inflammation and bleeding that perpetuate a disease-promoting ecosystem.

Oral hygiene is a daily personal protocol for effective delivery of active substances to the tissues of the oral cavity, mainly fluoride and antiseptics. The standard of care in the oral compound is toothpaste used 2-3 times a day.

The test toothpaste including Saliactive® (an olive product, betaine and xylitol) does not contain any antimicrobial agent nor antiseptic. A randomized, double-blind controlled clinical trial in 100 patients will evaluate the efficacy to reverse oral dysbiosis. Microbiota profile through genetic sequenciation of the rDNA16s, inflammatory markers, nitrate reducing bacteria abundance, nitrite/nitrate ratio, pH, plaque and bleeding index will be evaluated at baseline, after 2 months and 4 months of exposure to the assigned composition. Two controls will be analysed, one fluoridated placebo but without the 3 active ingredients olive product, betaine and xylitol (Saliactive®), and a fluoridated commercial toothpaste for gingivitis with zinc citrate. Assignation of the 100 subjects will be randomized and the products are blind for the subjects and the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose of gingivitis.
* At least 20 teeth (3rd molars excluded).
* Must Accept informed consent.

Exclusion Criteria:

* Clinical diagnose of periodontitis.
* With orthodontics.
* With removable dentures.
* With upper incisors restorated.
* Tumours in soft or hard tissues of the mouth.
* More than 5 caries lesions with immediate restorative need
* Antibiotics intake less than one month ago.
* Pregnant women.
* Other clinic assay at the moment.
* Dental prophylaxis less than 2 weeks before starting the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Oral microbiota profile at baseline and after 4 months | 4 months
  16s rDNA genetic sequencing
Oral pH at baseline and after 4 months | 4 months
  pH meter
Nitrite/Nitrate ratio at baseline and after 4 months | 4 months
  Ionic chromatography
Elastase at baseline at 2 months and at 4 months | 4 months
  ELISA
Bleeding index at baseline, at 2 months and at 4 months | 4 months
  Ainamo and Bay bleeding index indicating the percentage of bleeding from 0 (no bleeding) to 100 (maximum bleeding)
Plaque index at baseline, at 2 months and at 4 months | 4 months
  Tonetti plaque index

SECONDARY OUTCOMES:
Salivary flow rate at baseline, 2 months and at 4 months | 4 months
  Unstimulated salivary flow rate recovery as per Navazesh

OTHER OUTCOMES:
Tooth colour at baseline and at 4 months | 4 months
  VITA Easyshade® V

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Luis Mesa Aguado, Principal Investigator — Departamento de Estomatología, Facultad de Odontología
Locations (1):
- Departamento de Estomatología, Facultad de Odontología, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS. The future of periodontology: new treatments for a new era. J Int Acad Periodontol. 2002 Jul;4(3):110-4. PMID 12670090
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Navazesh M. Methods for collecting saliva. Ann N Y Acad Sci. 1993 Sep 20;694:72-7. doi: 10.1111/j.1749-6632.1993.tb18343.x. No abstract available. PMID 8215087
- [Background] Barbadoro P, Ponzio E, Coccia E, Prospero E, Santarelli A, Rappelli GGL, D'Errico MM. Association between hypertension, oral microbiome and salivary nitric oxide: A case-control study. Nitric Oxide. 2021 Jan 1;106:66-71. doi: 10.1016/j.niox.2020.11.002. Epub 2020 Nov 10. PMID 33186726
- [Background] Bescos R, Ashworth A, Clarke C, Brookes ZL, Belfield L, Rodiles A, Casas-Agustench P, Farnham G, Liddle L, Burleigh M, White D, Easton C, Hickson M. Effects of Chlorhexidine mouthwash on the oral microbiome. Sci Rep. 2020 Mar 24;10(1):5254. doi: 10.1038/s41598-020-61912-4. PMID 32210245